CLINICAL TRIAL: NCT03383250
Title: Factors to Determine the Responses to Meal Ingestion: Circulating Metabolites
Brief Title: Metabolomic Response to Meal Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR(AG)338/2016D
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: meal ingestion; postprandial sensations; circulating metabolites

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meal ingestion (Experimental)
  Interventions: Dietary Supplement: Normal meal

INTERVENTIONS:
Dietary Supplement: Normal meal

SUMMARY:
The investigators have recently shown that postprandial sensations correlate with changes in circulating metabolites after a meal ingestion; however this phenomenon was demonstrated with a meal load up to the level of tolerance which involved an unpleasant fullness sensation. The aim of the present study is to determine changes in circulating metabolites of a satiating pleasurable meal. Healthy men (n = 32) will be evaluated after a 5 h fast. Perception measurements and blood samples will be taken before and 20 minutes after ingestion of a palatable probe meal (juice and warm ham and cheese sandwich, total 300 ml, 440 kcal). NMR spectroscopy will be performed to determine plasmatic Low Molecular Weight Metabolites (LMWM) and to characterize lipoprotein profiles (number of particles, lipid content and size of the main three lipoprotein classes (VLDL, LDL and HDL). Homeostatic (satiety, fullness) and hedonic sensations (digestive well-being, mood) will be measured by 10 cm analogical scales.

ELIGIBILITY:
Inclusion Criteria:

* non obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Metabolomic response in serum | 30 min

SECONDARY OUTCOMES:
Change in digestive well-being measured after the test meal | 1 day
  Change in average well-being measured by 10 score scales at the end of the test meal.
Change in satiety measured after the test meal | 1 day
  Change in average satiety measured by 10 score scales at the end of the test meal
Change in fullness sensation measured after the test meal | 1 day
  Change in average fullness measured by 10 score scales at the end of the test meal
Change in abdominal discomfort/pain sensation measured after the test meal | 1 day
  Change in average abdominal discomfort/pain measured by 10 score scales at the end of the test meal
Change in mood measured after the test meal | 1 day
  Change in average mood measured by 10 score scales at the end of the test meal.